CLINICAL TRIAL: NCT06744283
Title: The Experience and Management of Cancer Screening-Related Anxiety in Fanconi Anemia: an Ethnographic Study
Brief Title: Experience and Management of Cancer Screening-Related Anxiety in Fanconi Anemia
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002289; 002289-C
Record Dates: First submitted 2024-12-19; First posted 2024-12-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-21

CONDITIONS: Fanconi Anemia
Keywords: Uncertainty; Fanconi Anemia; Cancer; Screening
MeSH Terms: conditions — Fanconi Anemia; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with a diagnosis of Fanconi anemia: Participants enrolled in the Fanconi Anemia Cancer Screening Study (FACSS) protocol (NIH IRB #: 001109) who are 18 years of age or older are eligible for inclusion in this study.

SUMMARY:
Background:

Fanconi anemia (FA) is a rare, inherited cancer syndrome. FA causes a range of physical issues. Children with FA may have abnormal features; these may include a small head and eyes and issues with their internal organs. Young adults have a much higher risk of cancer. To screen for these cancers, people with FA may need to pursue many visits with different doctors. This constant need for cancer screening may cause anxiety for people with FA.

Objective:

To learn more about anxiety related to cancer screenings in people with FA.

Eligibility:

Adults aged 18 years and older with FA. They must also be enrolled in FACSS. FACSS is a study that screens people with FA for cancer every year.

Design:

All data gathered for this study will occur during routine FACSS visits. No other visits are needed.

An observer will be in the room during participants FACSS visits. The observer and participant will have a polite introduction. After that, the observer will not interact with participants in any way.

The observer will note details about the participants, such as:

* Body language.
* Worries about screening.
* Comments that suggest anxiety or depression.
* Clinical environment, such as d(SqrRoot)(Copyright)cor and temperature.
* Accessibility issues. These can include lights and noises as well as ease of traveling around the clinic center.
* Evidence of social support, such as engaging in the FA community.
* Challenges they ve had in FACSS.
* Their motivation to participate in FACSS.
* Relationship dynamics among clinic staff, participants, and their care partners.

Data will also be collected from FACSS visit notes dating back to December 2024 and from participants medical records.

DETAILED DESCRIPTION:
Study Description:

This study will explore the experience and management of screening related anxiety in Fanconi Anemia (FA) among participants in the Fanconi Anemia Cancer Screening Study (FACSS) protocol (NIH IRB #:001109). Knowledge generated from this study will improve understanding of the experience and management of cancer screening-related anxiety in the context of complex, rare disease, while providing much-needed information about the health experiences and challenges within the FA community.

Objectives:

To collect ethnographic observational field notes to explore the nature of cancer screening-related anxiety experienced by participants in the FACSS screening study at the NIH clinical center.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants enrolled in the FACSS protocol who are 18 years of age or older are eligible for inclusion in this study. Clinical visits eligible for ethnographic observation are limited to initial visits (medical history and physical examination) and/or return of results visits happening in the context of their first visit to the NIH Clinical Center for the FACSS protocol and/or annual return visits.

To be eligible, the following requirements must be met:

* Ability for the participant to speak, read, and/or write in English to understand and agree to a verbal consent.
* Participants must have a diagnosis of FA.
* Participants must be 18 years of age or older.

EXCLUSION CRITERIA:

* Individuals who do not meet eligibility criteria.
* Subjects who declined or opted out of allowing their data to be used for future research.
* Subjects who orally declined to have Dr. Emily Pearce shadow their clinical center visits.
* No other exclusionary criteria apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study team will conduct a concurrent mixed methods study involving ethnographic data collected from field notes of clinical visits for participants in the Fanconi Anemia Cancer Screening Study (FACSS) protocol (NIH IRB #: 001109), including initial intake and/or return of results.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Examine screening-related anxiety usingethnographic field note | At Clinical Center Visit
  This mixed methods study will examine screening-related anxiety using ethnographic field notes include: 1) content analysis of predetermined categories of observation, and 2) qualitative analysis of field notes describing patient provider communication.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Savage, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Participants will not receive individual research results. Aggregate results of the research will be presented to the Fanconi Cancer Foundation (formerly Fanconi Anemia Research Fund) leadership and will be developed into a manuscript for publication.